CLINICAL TRIAL: NCT05186870
Title: A Study Investigating the Test- and Retest Reliability of a Battery of Functional Standardised Outcome Measures in Adults With Neurofibromatosis 1
Brief Title: Reliability of Functional Outcome Measures in Neurofibromatosis 1: Test- Retest
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 253954
Record Dates: First submitted 2021-03-23; First posted 2022-01-11 (Actual); Last update posted 2023-03-03 (Actual); Status verified 2023-03

CONDITIONS: Neurofibromatosis Type 1
MeSH Terms: conditions — Neurofibromatosis 1 | interventions — Outcome Assessment, Health Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Outcome measures — Observational study

SUMMARY:
To examine the test-retest reliability (how stable the results are when the same participants, whose symptoms have remained stable, are assessed on 2 different occasions, 14 days apart) of the 10 meter walk test, the timed up and go test, the functional reach test and the grip dynamometry test in adults with neurofibromatosis 1 (NF1).

DETAILED DESCRIPTION:
Participants' will be recruited during their attendance to the National Centre for Neurofibromatosis at Guy's hospital between August 2019 and March 2020 then following a COVID-19 break, from March 2022 until October 2022. Guy's and St Thomas' Trust (GSTT) is a National Centre for the diagnosis, management and support of approximately 1600 people with neurofibromatosis 1. Currently patients' attend the clinic for their standard assessment appointment every 6-12 months. They will receive a participant information sheet before their appointment, and the treating clinician (specialist doctors and nurses) will confirm that the individual meets the inclusion criteria and identify whether they wish to participate. At each of these contact points as well as within the participant information sheet, the potential participant will be advised that their decision to participate/ not to participate within this study will have no impact on their clinical care. Each participant will be asked to complete each outcome measure at both study visits.

Once written consent has been obtained each participant will be given a unique alphanumeric identification code for use within the trial. Written consent to participate in the study will be collected from the participant by the researcher (FD) on the day of their first outcome measure appointment. The researcher will then start the outcome measurement testing session. The participant will be expected to attend one additional appointments to their standard bi-yearly/yearly appointment where data on the outcome measure will only be collected, the additional appointment will be 14 days later. During each of these appointments the participants will be asked to complete 4 outcome measures (Timed-up and go, Timed 10m walk test, Functional reach test and Grip-A Dynamometry) 3 times (and a mean will be taken) alongside completion of the neurofibromatosis 1 quality of life questionnaire (INFQOL), and a basic neurological assessment (to establish a baseline of symptoms) During their second appointment, in addition to above, the participant will also be asked if they have noted any changes in their symptoms in the last 14 days. The testing procedure will take approximately 60 minutes per participant in total outside of the individual's clinic appointment time.

Outcome measures The 10m walk test will time how long it takes the participant to walk for a distance of 10m (this will be on a marked walkway). The timed up and go test will time how long it takes the participant to stand up from a chair, walk 3m, turn around and return to sitting on the chair. For each of the above tests the participant will complete them independently but can use a walking aid if they require to. The functional reach test will require the participant to stand with there arm out in front of them and reach forward as far as they can without moving their feet, the distance will be recorded with a tape measure attached to the wall. The final test, the grip dynamometry with require the participant to squeeze the Grip-A Dynamometer as hard as they can. They will complete these 3 times and a mean score will be taken.

Data Analysis and sample size Data will be collected and analyzed using Pearson and intra-class correlation models. These models are recommended when testing for reliability as repeated measurements cannot be regarded as randomized samples (Koo and Li, 2016). A sample of 20 (5 x the items to be tested) participants is recommended for use in test- retest studies (Park et al., 2017) to ensure that the sample is representative of the wider population. Once the data has been analyzed by the relevant clinician's the data will be destroyed in line with trust policy.

The researcher will not be involved in the initial invitation of participants to the study and will have no influence on who can join the study other than providing the inclusion and exclusion criteria. The participants overall standard care will not be affected through participation in the study inclusive if the recruitment process. In accordance with Good Clinical Practice (GCP) we will ensure that participants understand fully the reason for the study and their involvement.

Inclusion/exclusion criteria All participants aged 16 years or older who fulfill the diagnostic criteria for neurofibromatosis 1, who do not have a significant mobility or balance impairment that is unrelated to their neurofibromatosis 1, are able to walk more than 10 meters without physical assistance (may use walking aids), who are able to provide written consent and who attend the national Neurofibromatosis service at GSTT will be eligible to participate in the study.

Consent Participants will be recruited by the researcher (chief investigator) will obtain written consent to participate in the study a from every individual after they have had at least 24 hours to read the information sheet and the opportunity to ask questions about the study. Consent will be obtained by the chief investigator who has attended Good Clinical Practice Training.

Steps to reduce researcher bias To reduce the risk of selection bias, multiple clinicians will be included in recruitment however, the researcher will not be involved in this process.

To reduce the risk of performance bias, the outcome measurements will all be collected by the same Physiotherapist with standardized instructions.

To reduce the risk of detection bias, a statistician will review the statistical plan and the data collected to ensure appropriateness and accuracy.

ELIGIBILITY:
Inclusion Criteria:

* Patients who

  1. fulfill the diagnostic criteria for neurofibromatosis 1
  2. are aged 16 years or over
  3. attend the national neurofibromatosis service at GSTT
  4. are capable of providing informed consent
  5. do not have any non neurofibromatosis 1 related co-morbidities that affect mobility or balance (confirmed with the treating clinician)
  6. are able to walk more than 10 metres without assistance of a person (may use walking aid/orthotics)
  7. Symptoms that have remained stable between the 2 testing sessions (14 days). This will be assessed with the use of a neurological examination (Power, Sensation, Co-ordination, proprioception and reflexes), the NFQOL questionnaire and a subjective question to the patient as to if they feel there have been any changes to their symptoms in the last 14 days (completed on a percentage, 0= no change, 100% large change impacting their function). The assessing clinician will determine if any change is a significant change based on a reduction in power of more than 1 point (Oxford scale 0-5) and if there is a significant change in scores in comparison with the published norms.

Exclusion Criteria:

* Patients who

  1. do not fulfill the diagnostic criteria for neurofibromatosis 1
  2. are under the age of 16 years
  3. are unable to provide informed consent
  4. have non neurofibromatosis 1 related co-morbidities that affect mobility or balance (confirmed with the treating clinician)
  5. are unable to walk more than 10 metres without assistance of a person (may use walking aid/orthotics)
  6. Patients whose symptoms have not remained stable between the 2 testing sessions (14 days). This will be assessed with the use of a neurological examination (Power, Sensation, Co-ordination, proprioception and reflexes), the NFQOL questionnaire and a subjective question to the patient as to if they feel there have been any changes to their symptoms in the last 14 days (completed on a percentage, 0= no change, 100% large change impacting their function). The assessing clinician will determine if any change is a significant change based on The assessing clinician will determine if any change is a significant change based on a reduction in power of more than 1 point (Oxford scale 0-5) and if there is a significant change in scores in comparison with the published norms.
  7. If the participant has been involved in research which may impact the testing (e.g. changes in treatment which may impact their symptoms during the trial/currently involved in a study completing the same outcome measures and adding a level of learned bias) then they will not be invited to join the study.

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Participants' attending to the National Centre for Neurofibromatosis at Guy's hospital between August 2019- October 2019, January 2020-March 2020 and May 2022 until October 2022 then January 2023- June 2023. With extensions due to multiple issues during the trial recruitment periods including COVID and staffing change related.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2019-11-30 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Timed 10 meter walk test. | Baseline
  Time how long it takes the participant to walk for a distance of 10m
Timed 10 meter Walk test. | 14 days
  Time how long it takes the participant to walk for a distance of 10m
Timed up and Go | Baseline
  Time how long it takes the participant to stand up from a chair, walk 3m, turn around and return to sitting on the chair
Timed up and Go | 14 days
  Time how long it takes the participant to stand up from a chair, walk 3m, turn around and return to sitting on the chair
Functional reach test | Baseline
  Requires the participant to stand with there arm out in front of them and reach forward as far as they can without moving their feet, the distance will be recorded with a tape measure attached to the wall.
Functional reach test | 14 days
  Requires the participant to stand with there arm out in front of them and reach forward as far as they can without moving their feet, the distance will be recorded with a tape measure attached to the wall.
Grip dynamometry | Baseline
  Require the participant to squeeze the Grip-A Dynamometer as hard as they can. They will complete these 3 times and a mean score will be taken.
Grip dynamometry | 14 days
  Require the participant to squeeze the Grip-A Dynamometer as hard as they can. They will complete these 3 times and a mean score will be taken.

CONTACTS AND LOCATIONS:
Locations (1):
- Guy's Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No